CLINICAL TRIAL: NCT00000685
Title: Evaluation of Zidovudine Pharmacokinetics in Patients With Human Immunodeficiency Virus and Varying Degrees of Renal Insufficiency
Brief Title: A Study of Zidovudine in HIV-Infected Patients With Kidney Problems
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 088; NSC 602670; 11063 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-02 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Kidney Disease
Keywords: Kidney Diseases; Drug Evaluation; Acquired Immunodeficiency Syndrome; Zidovudine; Renal Dialysis
MeSH Terms: conditions — HIV Infections; Kidney Diseases; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine how zidovudine (AZT) for the treatment of HIV infection is metabolized and excreted or eliminated in patients with infected or diseased kidneys. To determine the influence of hemodialysis and establish dose guidelines.

AZT is the only antiviral agent with demonstrated effectiveness in patients with severe HIV infection. Persons with HIV infection may have additional health problems, one of which is a diseased kidney due to infection of the kidney, or side effects of therapy. The benefits and risks of AZT in patients with diseased kidneys are unknown. It is hoped that this study will allow further understanding of the metabolism and excretion of AZT in patients with kidney disease. AZT pharmacokinetics will be studied in patients with mild, moderate, and severe renal disorders

DETAILED DESCRIPTION:
AZT is the only antiviral agent with demonstrated effectiveness in patients with severe HIV infection. Persons with HIV infection may have additional health problems, one of which is a diseased kidney due to infection of the kidney, or side effects of therapy. The benefits and risks of AZT in patients with diseased kidneys are unknown. It is hoped that this study will allow further understanding of the metabolism and excretion of AZT in patients with kidney disease. AZT pharmacokinetics will be studied in patients with mild, moderate, and severe renal disorders.

Patients receive AZT by mouth on the first day. After taking the AZT, blood samples are taken from a catheter and several urine samples are collected over a 24-hour period. During this time, patients remain in the hospital for the 24 hours or may choose to go home 12 hours after taking the AZT dose and return for the last blood sample the next morning. Following study day 1, patients receive AZT every 4 hours, including in the middle of the night, and keep a diary of the times they take AZT, as well as of the use of other medications, tobacco, or alcohol. A return appointment is made for 8-15 days later. On that day, patients again receive AZT by mouth, and blood tests and urine samples are again taken. Patients who are receiving hemodialysis participate in 1 additional day of pharmacokinetic studies to be arranged during one hemodialysis session. Patients on Continuous Ambulatory Peritoneal Dialysis (CAPD) are studied separately and do not participate in the procedures for the other groups. AZT is given as a single oral dose at the beginning of the first morning exchange followed by a pharmacokinetic study. Chronic AZT dosing is initiated following the first exchange. After a minimum of 7 days of AZT therapy and a maximum of 14 days the last dose of AZT is administered and a repeat pharmacokinetic study is done. All patients are seen again 1-2 weeks after completing the last pharmacokinetic study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Symptomatic therapy such as analgesics, antihistamines, antiemetics, antidiarrheal agents, or other supportive therapy.
* Aerosolized pentamidine.

Discouraged:

- Sucralfate or antacids. However if these medications are essential for the patient's management, they should not be given within 8 hours before or 2 hours after the scheduled pharmacokinetic study.

-

Concurrent Treatment:

Allowed:

* Blood transfusions.

Patients must have HIV infection with renal insufficiency and acceptable hepatic and hematologic function. They must have been on dialysis treatment for at least 3 months.

Prior Medication:

Allowed:

* Cytotoxic chemotherapy for local mucocutaneous lesions.
* Aerosolized pentamidine.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Ongoing therapy for opportunistic infections, including systemic maintenance therapy which cannot be discontinued for the duration of the study, such as amphotericin B or ganciclovir.
* H-2 blockers.
* Zidovudine (AZT).
* Other antiretroviral agents or other experimental therapy.

Discouraged:

- Sucralfate or antacids. However, if these medications are essential for the patient's management, they should not be given within 8 hours before or 2 hours after the scheduled pharmacokinetic study.

-

Patients will be excluded from the study for the following reasons:

* Presence of active opportunistic infections.
* Severe malabsorption syndrome (persistent diarrhea greater than 4 weeks duration with = or > 4 loose stools per day accompanied by = or > 10 percent unintentional weight loss.
* Acute illness, febrile or unstable, 48 hours prior to the first pharmacokinetic study.
* Known sensitivity to zidovudine or thymidine-type agents.
* Diabetes mellitus requiring treatment.

Prior Medication:

Excluded:

- Treatment for diabetes mellitus.

Excluded within 72 hours of study entry:

* H-2 blockers.
* Zidovudine (AZT).

Excluded within 2 weeks of study entry:

* Other antiretroviral agents or other experimental therapy.
* Rifampin or rifampin derivatives.
* Probenecid.
* Dilantin.
* Methadone.
* Oral contraceptives.
* Barbiturates.
* Significant hepatotoxic agents or valproic acid.
* TMP / SMX.
* Dapsone.
* Fansidar.

Excluded within 30 days of study entry:

- Cytotoxic chemotherapy.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy for local mucocutaneous lesions.

Risk Behavior:

Active drug or alcohol use which might interfere with the study objectives.

* Note: Alcohol consumption is prohibited 48 hours prior to the first pharmacokinetic study and during the study. Tobacco smoking is not excluded although tobacco use will be quantified.

Patients may not have any of the following diseases or symptoms:

* Presence of active opportunistic infections.
* Severe malabsorption syndrome (persistent diarrhea greater than 4 weeks duration with = or > 4 loose stools per day accompanied by = or > 10 percent unintentional weight loss.
* Acute illness, febrile or unstable, 48 hours prior to the first pharmacokinetic study.
* Diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tartaglione TA, Study Chair
Locations (2):
- United States (2):
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Tartaglione TA, Holeman E, Opheim K, Smith T, Collier AC. Zidovudine disposition during hemodialysis in a patient with acquired immunodeficiency syndrome. J Acquir Immune Defic Syndr (1988). 1990;3(1):32-4. PMID 2293640